CLINICAL TRIAL: NCT06904261
Title: An Open-label Study of the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of 12 Month Treatment With Migalastat in Pediatric Subjects (Aged 2 to < 12 Years) With Fabry Disease and Amenable GLA Variants
Brief Title: A Study of Migalastat in Pediatric Subjects (2 to <12 Yrs) With Fabry Disease and Amenable GLA Variants
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amicus Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT1001-033
Expanded Access: NCT01476163 (Available)
Record Dates: First submitted 2025-03-13; First posted 2025-04-01 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-06

CONDITIONS: Fabry Disease
Keywords: migalastat; AT1001; Galafold; lysosomal disease
MeSH Terms: conditions — Fabry Disease | interventions — migalastat; larazotide acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Migalastat HCl 20 mg Dispersible Tablets (Experimental): Migalastat will be administered every other day (QOD). The initial dose will be based on body weight at baseline.
  Interventions: Drug: Migalastat HCl 20 mg

INTERVENTIONS:
Drug: Migalastat HCl 20 mg — Migalastat will be supplied as 20-mg dispersible tablets. Migalastat 20-mg dispersible tablets contain 16 mg migalastat free base.
  Other Names: AT1001; Galafold

SUMMARY:
An open-label study to evaluate the safety, pharmacokinetics (PK), pharmacodynamics (PD), and efficacy of migalastat treatment in pediatric subjects 2 to < 12 years of age with Fabry disease and with amenable GLA variants.

DETAILED DESCRIPTION:
This is a Phase 3b, 2-stage, open-label, uncontrolled, multicenter study to evaluate the safety, PK, PD, and efficacy of 12 months of migalastat treatment in pediatric subjects 2 to < 12 years of age with Fabry disease and with amenable GLA variants. Subjects must be either naïve to enzyme replacement therapy (ERT) or have stopped ERT at least 14 days before Baseline visit.

The study will consist of 2 treatment stages followed by an open-label extension (OLE). Stage 1 will be a treatment period of approximately 3 months (12 weeks); Stage 2 will be a treatment period of 9 months. There will be no break in treatment between Stages 1 and 2. There will be a 30-day (untreated) safety follow-up period for subjects who discontinue treatment at any time.

Subjects will be randomly assigned 1:1:1 to 1 of 3 PK sampling groups using interactive response technology (IRT). Four blood samples for the determination of migalastat concentrations in plasma will be collected in one 24-hour period between Day 15 and Day 30 and at Month 6, and 1 PK (trough) sample will be collected at Month 6 and again at Month 12.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects, diagnosed with Fabry disease who are between ages 2 and < 12 years at randomization (subjects aged 11 years must have birthdays > 30 days after randomization)
* Subject's parent or legally authorized representative is willing and able to provide written informed consent and authorization for use and disclosure of personal health information or research-related health information, and subject provides assent, if applicable.
* Subject has a GLA variant documented in his/her medical record that is amenable to migalastat prior to Visit 2.
* Subject has not received ERT (eg, Replagal® [agalsidase alfa] or Fabrazyme® [agalsidase beta]) for at least 14 days prior to Baseline visit.
* Subject has at least 1 documented complication (ie, historical or current laboratory abnormality or sign/symptom) of Fabry disease
* If of reproductive potential, both male and female subjects agree to use a medically accepted method of contraception throughout the duration of the study and for up to 30 days after their last dose of migalastat.

Exclusion Criteria

* Has moderate or severe renal impairment (eGFR < 60 mL/min/1.73 m2 at Visit 1 [screening]).
* Has advanced kidney disease requiring dialysis or kidney transplantation.
* History of allergy or sensitivity to migalastat (including excipients) or other iminosugars (eg, miglustat, miglitol).
* Has received any investigational/experimental drug, biologic, or device within 30 days or 5 half-lives of the investigational product (whichever is longer) before Visit 1 (screening).
* Has received any gene therapy at any time or anticipates starting gene therapy during the study period.
* Requires treatment with Glyset (miglitol) or Zavesca (miglustat), within 6 months before Visit 1(screening) or throughout the study.
* Has any intercurrent illness or condition at Visit 1 (screening) or Visit 2 (baseline) that may preclude the subject from fulfilling the protocol requirements or suggests to the investigator that the potential subject may have an unacceptable risk by participating in this study.
* Pregnant or breastfeeding
* Otherwise unsuitable for the study in the opinion of the investigator

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Safety: Incidence of TEAEs, SAEs, and AEs leading to discontinuation of study drug | Day 1 (after dosing) through Month 12 and follow-up (30 days after last dose)
Pharmacokinetics (PK): Maximum Observed Plasma Concentration (Cmax) of Migalastat | 0 to 12 hours postdose during the first month of study and trough samples at Months 6 and 12
Pharmacokinetics (PK): Minimum Observed Plasma Concentration (Cmin) of Migalastat | 0 to 12 hours postdose during the first month of study and trough samples at Months 6 and 12
Pharmacokinetics (PK): Area Under The Plasma Concentration-time Curve Over The Dosing Interval (AUCtau) of Migalastat | 0 to 12 hours postdose during the first month of study and trough samples at Months 6 and 12

SECONDARY OUTCOMES:
Pharmacodynamic: Change in plasma levels of lyso-Gb3 and its analogs from baseline | Baseline to Months 3, 6, and 12/ET
Efficacy: Change in eGFR from baseline | Baseline to Months 1, 3, 6, and 12/ET
  eGFR is calculated using the modified Schwartz formula for creatinine clearance. eGFR will also be calculated separately using the CKD-EPI40 equation.
Efficacy: Change in urine protein and albumin/microalbumin levels from baseline | Baseline to Months 3, 6, and 12/ET
Efficacy: Change in Left Ventricular Mass Index (LVMi) from baseline | Baseline to Month 12/ET
Efficacy: Change in FABPRO-GI And Pain Scores from baseline | Baseline to Month 12/ET
  The Fabry Disease Patient-Reported Outcome - Gastrointestinal Signs And Symptoms (FABPRO-GI) And Pain Questionnaire For Clinical Trials (24-hr Version) consists of questions regarding gastrointestinal signs and symptoms and pain relative to the past 24 hours. Participants rate the severity of their symptoms and pain from 0 (none) to 10 (worst possible). A higher score indicated higher levels of symptoms and pain.
Efficacy: Mean Patient's Global Impression Of Change (PGI-C) values | Months 3, 6, and 12/ET
  The PGI-C consists of 4 questions regarding diarrhea, abdominal pain, overall pain, and daily living. Participants rate their status based on improvement, worsening, or the same. Improved status includes "Much better", "Better" and "A little better"; worsened status includes "A little worse", "Worse" and "Much worse".
Efficacy: Change in EQ-5D-Y scores from baseline (subjects aged ≥4 years) | Baseline to Month 12/ET
  The EuroQol 5-dimension Youth Questionnaire [EQ-5D-Y] is a two-part instrument: the EQ-5D descriptive system and the EQ visual analogue scale (VAS). The descriptive system covers five health domains: mobility, looking after myself, doing usual activities, having pain or discomfort and feeling worried, sad or unhappy. Each domain has 3 response categories: no problems, some problems and a lot of problems. The response categories can be reflected by a 1-digit number (1-3) and combined for the five dimensions into a 5-digit number to describe the health state of the patient. The EQ VAS records the patient's self-rated health on a vertical VAS of 0-100 where 100="The best health you can imagine" and 0="The worst health you can imagine". The VAS can be used as a quantitative measure of health outcome that reflects the patient's own judgement.
Efficacy: Change in PedsQL scores from baseline | Baseline to Month 12/ET
  The Pediatric Quality of Life Inventory™ (PedsQL) is a modular approach to measuring health-related quality of life in healthy children and adolescents and those with acute and chronic health conditions. The psychosocial score for the PedsQL encompasses 15 questions relating to the participants' feelings, social interaction with others, and school. The physical score is derived from answers to 8 questions about the participants' ease of managing physical activity. All components of the PedsQL are scored based on a scale of 0 (never) to 4 (almost always) and linearly transformed to a 0-100 scale as follows: 0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0. Both categories are combined for a total score.
Efficacy: Change in FPHPQ scores from baseline (subjects aged ≥4 years) | Baseline to Month 12/ET
  The Fabry-specific Pediatric Health and Pain Questionnaire (FPHPQ) includes questions about Fabry disease-specific symptoms (eg, sweating, pain, dizziness and tiredness, heat and cold intolerance, swollen eyelids, gastrointestinal symptoms, feeling thirsty, difficulty hearing, ringing or buzzing noise in the ears, and ability and enjoyment to participate in sports). The frequency of these symptoms will be rated using a 5-point Likert scale (always, often, sometimes, seldom, never). Pain intensity is measured on a 10-point scale with numeric responses given for onset of pain and school days missed, and yes/no questions posed about difficulty hearing and other problems not specifically mentioned.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (4):
  - Emory Genetics, Atlanta, Georgia
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Lysosomal and Rare Disorders Research and Treatment Center, Inc., Fairfax, Virginia
- Universitair Ziekenhuis (UZ) Leuven, Leuven, Vlaams-Brabant, Belgium
- Universitäetsklinikum Müenster (UKM) Klinik für Kinder- und Jugendmedizin - Allgemeine Paediatrie, Münster, North Rhine-Westphalia, Germany
- Hospital Universitario de la Paz, Madrid, Madrid, Spain
- United Kingdom (2):
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Undecided
Data sharing proposals and requests will be reviewed on a case-by-case basis. Requests for data should be addressed to Nick Rees at nrees@amicusrx.com. Requests will be reviewed by a medical steering committee.